CLINICAL TRIAL: NCT07225738
Title: A Multicenter Prospective Observational Cohort Study Evaluating the Impact of Cancer-Directed Treatment and Medication Use, Including Cannabis Use, in Multiple Myeloma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 25077; NCI-2025-07334 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25077 (Other: City of Hope Medical Center); P30CA033572 (NIH); U01CA286808 (NIH)
Record Dates: First submitted 2025-10-16; First posted 2025-11-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational group I: Patients complete surveys and undergo blood sample collection throughout the study.
  Interventions: Other: Non-Interventional Study
- Observational group II: Healthcare providers complete a survey on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
This study assesses the impact of cannabis (also commonly called marijuana, weed, or THC) use on quality of life among patients with multiple myeloma who are receiving chemotherapy. It also evaluates the potential benefits and harms of cannabis use.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Characterize and compare longitudinal patterns in quality of life, as assessed by the Functional Assessment of Cancer Therapy-Multiple Myeloma (FACT-MM) instrument, among cannabis users and non-users.

II. Estimate and characterize the potential therapeutic benefit and adverse effects associated with cannabis use as assessed by longitudinal patterns of patient reported symptoms (Edmonton Symptoms Assessment Scale-ESAS) and medical assessments (Common Terminology Criteria for Adverse Events-CTCAE v5.0) through a comparative analysis of users and non-users.

OUTLINE: This is an observational study. Participants are assigned to 1 of 2 groups.

GROUP I: Patients complete surveys and undergo blood sample collection throughout the study.

GROUP II: Healthcare providers complete a survey on study.

ELIGIBILITY:
Inclusion Criteria:

* * Documented informed consent of the participant

  * Age: ≥ 18 years
  * ECOG ≤ 3
  * Ability to read and understand English
  * Patient must be newly diagnosed with a histologically confirmed multiple myeloma
  * Patients may have started first line therapies and received up to four cycles
  * HCP SURVEY: Documented informed consent of the participant
  * HCP SURVEY: Age: ≥ 18 years
  * HCP SURVEY: Licensed physician, physician assistant, nurse practitioner, or registered nurse
  * HCP SURVEY: Currently practicing in oncology or providing direct care to oncology patients
  * HCP SURVEY: Able to read and understand English
  * HCP SURVEY: Affiliation with City of Hope

Exclusion Criteria:

* * Patients may not have completed five cycles of first line therapy or undergone any second line therapy

  * Other active malignancy
  * Patients may not have undergone autologous hematopoietic stem cell transplantation
  * Unable to comply with the study assessments
  * HCP SURVEY: Reports directly to study PI (Dr. Richard Lee)
  * HCP SURVEY: Member of the study team or involved in survey design or analysis
  * HCP SURVEY: Individuals with a real or perceived conflict of interest that could bias survey responses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed multiple myeloma patients who have received up to four cycles of first line therapy and City of Hope affiliated health care providers currently practicing in oncology or providing direct care to oncology patients.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-12-24 (Estimated); Primary Completion 2027-05-13 (Estimated); Study Completion 2027-05-13 (Estimated)

PRIMARY OUTCOMES:
Longitudinal patterns in quality of life | Up to one year
  Will characterize and compare longitudinal patterns in quality of life, as assessed by the Functional Assessment of Cancer Therapy-Multiple Myeloma (FACT-MM) instrument, among cannabis users and non-users. The analysis will compare difference scores from the FACT-MM between these groups using ANOVA at the end of treatment. For comparisons between groups at four specific assessment points (baseline, C1, C2, C3, and C4), a repeated measures analysis of variance analysis will be performed. Multivariable mixed-effects regression model, which takes possible dependence of longitudinal measurements within each subject into account, will be used. The possible within-subject dependence will also be taken into account using the robust standard error (generalized estimating equation method) when statistical inferences are made with regards to the treatment effect and interaction between treatment and time period.
Potential therapeutic benefit and adverse effects associated with cannabis use | Up to one year
  Will estimate and characterize the potential therapeutic benefit and adverse effects associated with cannabis use as assessed by longitudinal patterns of patient reported symptoms (Edmonton Symptoms Assessment Scale-ESAS) through a comparative analysis of users and non-users. Descriptive statistics will be computed regarding reported benefits and harms of cannabis, and associations will be explored with the different type of cannabis utilized.
Potential therapeutic benefit and adverse effects associated with cannabis use | Up to one year
  Will estimate and characterize the potential therapeutic benefit and adverse effects associated with cannabis use as assessed by medical assessments (Common Terminology Criteria for Adverse Events-CTCAE v5.0) through a comparative analysis of users and non-users. Descriptive statistics will be computed regarding reported benefits and harms of cannabis, and associations will be explored with the different type of cannabis utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Lee, Principal Investigator — City of Hope Medical Center
Locations (11):
- United States (11):
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - City of Hope Medical Center, Duarte, California
  - City of Hope Seacliff, Huntington Beach, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope at Long Beach Elm, Long Beach, California
  - City of Hope at Newport Beach Fashion Island, Newport Beach, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope Upland, Upland, California
  - City of Hope West Covina, West Covina, California
  - City of Hope Atlanta Cancer Center, Newnan, Georgia
  - City of Hope at Chicago, Zion, Illinois